CLINICAL TRIAL: NCT02963896
Title: Vertigo Perception and Quality of Life in Patients After Surgical Treatment of Vestibular Schwannoma With Pretreatment Prehabituation by Chemical Vestibular Ablation
Brief Title: Vertigo Perception and Quality of Life in Patients After Surgical Treatment of Vestibular Schwannoma
Acronym: ITG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Zdeněk Čada, M.D., PH.D., University Hospital, Motol
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13476 FN Motol
Record Dates: First submitted 2016-11-01; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Vestibular Schwannoma
Keywords: vestibular rehabilitation
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gentamicin (Experimental): intratympanic application of gentamicin 0.5 ml
  Interventions: Drug: gentamicin

INTERVENTIONS:
Drug: gentamicin — intratympanic application of gentamicin 2m/80mg - 3x application -0,5 ml
  Other Names: gentamycin

SUMMARY:
Surgical removal of vestibular schwannoma causes acute vestibular symptoms, including postoperative vertigo and oscilopsia due to nystagmus. In general, the dominant symptom postoperatively is vertigo. Preoperative chemical vestibular ablation can reduce vestibular symptoms postoperatively.

DETAILED DESCRIPTION:
Surgical removal of vestibular schwannoma causes acute vestibular symptoms, including postoperative vertigo and oscilopsia due to nystagmus. In general, the dominant symptom postoperatively is vertigo. Preoperative chemical vestibular ablation can reduce vestibular symptoms postoperatively. We used 1.0 ml of 40 mg/ml nonbuffered gentamicin in three intratympanic installations over 2 days, 2 months preoperatively in 10 patients. Reduction of vestibular function was measured by the head impulse test and the caloric test. Reduction of vestibular function was found in all gentamicin patient groups. After gentamicin vestibular ablation, patients underwent home vestibular exercising for two months. The control group consisted of 10 patients who underwent only home vestibular training two months preoperatively. Postoperative rate of recovery and vertigo in both groups were evaluated with the Glasgow Benefit Inventory (GBI), the Glasgow Health Status Inventory (GHSI) and the Dizziness Handicap Inventory questionnaires, as well as survey of visual symptoms by specific questionnaire developed by us.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of vestibular schwannoma
* hearing loss on affected side
* preserved vestibular reactivity of labyrinths on the affected side

Exclusion Criteria:

* allergy to gentamicin
* vestibular areflexia on the affected side

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The GBI questionnaire | 2-3 years
  The GBI questionnaire consists of 18 questions. The response to each question is based on a five-point Likert scale, ranging from a large deterioration to a large improvement in health status. The GBI questionnaire is scored into a total score, and also three subscales: a general subscale (12 questions), a social support subscale (three questions), and a physical health subscale (three questions). Score ranges were calculated and varied from -100 to +100. Score all questions so that a score of 1 is given to the answer with the worst change in health status and 5 to the answer with the best change in health status.
The GHSI questionnaire | 2-3 years
  The GHSI questionnaire contains of 18 questions; again, the response to each question is based on a five-point Likert scale ranging from high to low health status. It is also scored into a total score and three subscales: general, social, and physical health subscales. All these scores range from 0 to +100. Score all questions so that a score of 1 is given to the answer with the worst change in health status and 5 to the answer with the best change in health status.
The DHI questionnaire | 2-3 years
  The DHI contains 25 items and the range score is from 0 to +100, with a higher score indicating a more severe handicap.

CONTACTS AND LOCATIONS:
Overall Officials: Zdeněk Čada, Ph.D., Principal Investigator — Department of Otorhinolaryngology and Head and Neck Surgery, 1st Faculty of Medicine Charles University in Prague and Motol University Hospital, Postgraduate Medical School

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herdman SJ, Clendaniel RA, Mattox DE, Holliday MJ, Niparko JK. Vestibular adaptation exercises and recovery: acute stage after acoustic neuroma resection. Otolaryngol Head Neck Surg. 1995 Jul;113(1):77-87. doi: 10.1016/s0194-5998(95)70148-6. PMID 7603726
- [Derived] Cada Z, Balatkova Z, Chovanec M, Cakrt O, Hruba S, Jerabek J, Zverina E, Profant O, Fik Z, Komarc M, Betka J, Kluh J, Cerny R. Vertigo Perception and Quality of Life in Patients after Surgical Treatment of Vestibular Schwannoma with Pretreatment Prehabituation by Chemical Vestibular Ablation. Biomed Res Int. 2016;2016:6767216. doi: 10.1155/2016/6767216. Epub 2016 Dec 8. PMID 28053986